CLINICAL TRIAL: NCT02950701
Title: Data During Emergency Medical Transport in Suspected Carbon Monoxide Poisoning
Brief Title: Suspected Cases of Carbon Monoxide Poisoning
Status: Completed | Type: Observational
Sponsor: Nonin Medical, Inc (Industry)
Responsible Party: Sponsor
Other Study IDs: QATP2996
Record Dates: First submitted 2016-10-28; First posted 2016-11-01 (Estimated); Last update posted 2018-06-26 (Actual); Status verified 2016-10

CONDITIONS: Carbon Monoxide Intoxication
MeSH Terms: conditions — Carbon Monoxide Poisoning

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Device: Observational data collection.

SUMMARY:
The purpose of this study is to collect non-invasive opportunity sample data in suspected or known cases of carbon monoxide poisoning.

ELIGIBILITY:
Inclusion Criteria:

* Known or suspected carbon monoxide poisoning.

Exclusion Criteria:

* Less than 18 years of age

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The participants will be selected based on symptoms during medical transport.
Sampling Method: Non-Probability Sample
Enrollment: 82 (Actual)
Dates: Start 2016-11; Primary Completion 2017-09-22 (Actual); Study Completion 2017-09-22 (Actual)

PRIMARY OUTCOMES:
Values from the test device will be compared to the values from the reference device. | Through study completion, an average of 1 year.

CONTACTS AND LOCATIONS:
Overall Officials: Keith Wesley, MD, Principal Investigator — HealthEast Medical Transport
Locations (1):
- HealthEast Medical Transportation, Saint Paul, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No